CLINICAL TRIAL: NCT01701037
Title: Biomarkers of Response and Resistance to Sequential B-RAF and MEK Targeted Therapy in a Pre-Surgical Model of Advanced, Operable Melanoma
Brief Title: Dabrafenib Alone and in Combination With Trametinib Before Surgery in Treating Patients With Locally or Regionally Advanced Melanoma That Can Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI leaving VICC, low future accrual predicted, continued funding improbable,
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Mark Kelley, MD, Chief, Division of Surgical Oncology and Endocrine Surgery; Associate Professor of Surgery; Surgical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VICC MEL 1263; NCI-2012-01699 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-09-21; First posted 2012-10-04 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Recurrent Melanoma; Stage IIB Melanoma (Locally Advanced); Stage IIC Melanoma (Locally Advanced); Stage IIIA Melanoma; Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Melanoma (Limited, Resectable)
Keywords: Melanoma, B-RAF, biomarkers, targeted therapy, resistance
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dabrafenib and Trametinib (Experimental): Patients receive dabrafenib PO BID on days 1-28 adding trametinib on days 15-28 followed by surgery on days 28-30. Treatment continues in the absence of unacceptable toxicity.
  Interventions: Drug: dabrafenib; Drug: trametinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: dabrafenib — 150 mg given PO
  Other Names: BRAF inhibitor GSK2118436; GSK2118436
Drug: trametinib — 2 mg given PO
  Other Names: GSK1120212
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving dabrafenib alone and in combination with trametinib before surgery works in treating patients with advanced melanoma that can be removed by surgery. Studying samples of tumor tissue in the laboratory from patients receiving dabrafenib and trametinib may help doctors learn more about the effects of these drugs on cells and help identify biomarkers that determine which patients will respond to these drugs best.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify markers of intrinsic resistance to v-Raf murine sarcoma viral oncogene homolog B1 (B-RAF) targeted therapy in B-RAF mutation-positive melanoma.

SECONDARY OBJECTIVES:

I. To determine if intrinsic resistance can be reversed by mitogen activated protein kinase (MEK) targeted therapy and to identify biomarkers that correlate with this response.

II. To evaluate the feasibility of pre-surgical targeted therapy and serial tumor biopsies in patients with advanced, operable melanoma to determine if this model can be used to evaluate novel combinations of molecular targeted therapy in the future.

TERTIARY OBJECTIVES:

I. To determine if pre-surgical B-RAF and MEK targeted therapy is active and well tolerated in patients with advanced, operable melanoma. These findings may be used to support clinical trials in un-resectable, B-RAF mutation-positive melanoma.

OUTLINE:

Patients receive dabrafenib orally (PO) twice daily (BID) on days 1-28 adding trametinib on days 15-28 followed by surgery on days 28-30. Treatment continues until the day prior to surgery in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Patients with locally-or regionally advanced melanoma being considered for resection of the lesion(s) for local-regional control and potential cure

  * Patients with limited, resectable metastatic disease (three or fewer lesions) are eligible if surgical resection is considered to be the best therapeutic option
  * Patients with AJCC clinical stage IIb-IV disease at initial diagnosis, or patients with melanoma of any stage with advanced local or regional recurrence, with or without limited resectable metastatic disease, would be eligible
* B-RAF V-600 mutation positive by snapshot molecular analysis

  * Individuals with B-RAF V-600 mutations other than V600E are eligible
* Measurable disease, i.e. presenting with at least one measurable lesion per Response Evaluation Criteria in Solid tumors (RECIST) 1.1
* All prior treatment related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) (Version 4.0) =< Grade 1 at the time of enrollment
* Adequate baseline organ function defined by the criteria below:

  * Absolute Neutrophil Count (ANC) >= 1.5 X 10^9/L
  * Platelet Count >= 60 X 10^9/L
  * Hemoglobin >= 9 g/dl
  * Creatinine =< 2 mg/dl
  * Aspartate aminotransferase (AST) =< 100 U/L
  * Alanine aminotransferase (ALT) =< 100 U/L
  * Alkaline Phosphatase =< 380 U/L
  * Total Bilirubin =< 2.0 mg/dl
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of first dose of study treatment and agree to use effective contraception during the study and for 7 days following the last dose of study treatment
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from 1 day prior to administration of the first dose of study treatment until 7 days after the last dose of study treatment

Exclusion Criteria:

* ECOG Performance Status > 2
* Lactating female
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
* Any serious medical condition that would render the patient unable to undergo surgical resection or would limit life expectancy to less than 1 year
* Any prohibited medication
* Administration of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study treatment
* A known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to GSK-2118436 (dabrafenib) or GSK-1120212 (trametinib) or excipient that contraindicates their participation
* Patients with a history of severe cardiovascular disease as defined:

  * Symptomatic or uncontrolled cardiac arrhythmias
  * Treatment refractory hypertension, defined as a systolic blood pressure > 160mm Hg and/or diastolic > 100 mmHg which cannot be controlled by antihypertensive therapy.
  * Current ≥ NYHA Class II congestive heart failure
  * History of myocardial infarction or unstable angina within 6 months prior to study entry.
  * History of stroke or TIA within 6 months prior to study entry
  * QTc ≥ 480 msec
  * Cardiac valvular disease ≥ grade 2.
* Patients with a history of interstitial lung disease or interstitial pneumonitis
* A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection.
* History of another active malignancy within the past 5 years, or any malignancy with a confirmed activating RAS mutation. Please note that prospective RAS mutation testing is not required, however, if results of previous RAS testing are known, they must be used in assessing eligibility. Subjects with a history of completely resected non-melanoma skin cancer are eligible.
* A history or current evidence/risk of retinal vein occlusion (RVO) or CSR including:
* a. Presence of predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes); or
* b. Visible retinal pathology as assessed by ophthalmic examination that is considered a risk factor for RVO or CSR such as:

  * i. Evidence of new optic disc cupping;
  * ii. Evidence of new visual field defects on automated perimetry;
  * iii. Intraocular pressure >21 mmHg as measured by tonography.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-01; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kelley, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Johnson AS, Crandall H, Dahlman K, Kelley MC. Preliminary results from a prospective trial of preoperative combined BRAF and MEK-targeted therapy in advanced BRAF mutation-positive melanoma. J Am Coll Surg. 2015 Apr;220(4):581-93.e1. doi: 10.1016/j.jamcollsurg.2014.12.057. Epub 2015 Jan 30. PMID 25797743
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened to accrual at Vanderbilt-Ingram Cancer Center (VICC) in January 2013 and ran through March 2015 when it closed prematurely due to PI's departure.
Pre-assignment Details: Thirteen patients participated in this study, all completed the study as defined by protocol.
Groups:
- Basic Science (Dabrafenib, Trametinib): Patients receive dabrafenib PO BID on days 1-28 adding trametinib on days 15-28 followed by surgery on days 28-30. Treatment continues in the absence of unacceptable toxicity.
  dabrafenib: 150 mg given PO
  trametinib: 2 mg given PO
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Basic Science (Dabrafenib, Trametinib)
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Basic Science (Dabrafenib, Trametinib)
Number analyzed (Participants) | 13
Age, Customized [Count of Participants; unit: Participants]
  20-29 | 1
  30-39 | 2
  40-49 | 2
  50-59 | 3
  60-69 | 3
  70-79 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Clinical Tumor Response Rate (Response is Based on Greater Than 30% Reduction From Baseline in Tumor Volume by RECIST Criteria) at Day 14.
Description: Tumor response is defined as greater than 30% reduction from baseline in tumor volume by RECIST criteria. To determine whether a patient is responded at day 14, the patient must have the tumor volume evaluated at both baseline and day 14. The tumor response rate is calculated as the proportion of patients responded among all evaluated patients.
Time Frame: day 14
Measure: Number (95% Confidence Interval); unit: proportion of responders
Arm/Group | Dabrafenib and Trametinib
Number analyzed (Participants) | 12
proportion of responders | 0.833 [0.552 to 0.953]

2. Secondary Outcome: Change in Tumor Volume Reduction in Participants With Intrinsic Resistance to B-RAF Targeted Therapy From Day 14 to Day 28.
Description: Tumor volume reduction is calculated as the tumor volume change relative to the baseline measurement (percent). Change in tumor volume reduction from day 14 to day 28 is calculated as the difference of tumor volume reduction at day 28 and day 14. The median and Inter-Quartile Range are reported.
Time Frame: Day 14 and day 28
Measure: Median (Inter-Quartile Range); unit: percentage of reduction
Arm/Group | Dabrafenib and Trametinib
Number analyzed (Participants) | 11
percentage of reduction | 18.0 [16.5 to 23.5]

3. Secondary Outcome: Number of Patients With Worst Grade Toxicities by Grade According to National Cancer Institute (NCI) CTCAE Version 4.0
Description: The intensity of the adverse event will be graded according to Version 4.0 of the National Cancer Institute Common Terminology Criteria for Adverse Events (June 14, 2010):
  Grade 1 - Mild Grade 2 - Moderate Grade 3 - Severe or medically significant Grade 4 - Life-threatening Grade 5 - Death related to adverse event
Time Frame: Up to 3 months
Measure: Number; unit: participants
Arm/Group | Dabrafenib and Trametinib
Number analyzed (Participants) | 13
participants
  Number of patients with worst-grade toxicity 1 | 1
  Number of patients with worst-grade toxicity 2 | 6
  Number of patients with worst-grade toxicity 3 | 6
  Number of patients with worst-grade toxicity 4 | 0
  Number of patients with worst-grade toxicity 5 | 0

4. Secondary Outcome: Investigational Agent Taken
Description: Median number of pills taken
Time Frame: Up to 3 months
Measure: Median (Standard Deviation); unit: Number of pills taken
Arm/Group | Dabrafenib and Trametinib
Number analyzed (Participants) | 13
Number of pills taken
  Median number of GSK1120212 taken | 13 (1.90)
  Median number of GSK2118436 taken | 54 (6.34)

5. Secondary Outcome: Percent of Patients Completing Second and Third (Surgical) Biopsies
Description: Biopsies will be assessed whether or not tissue is acquired at specified time points. Tissue is obtained through core, punch, incisional or excisional biopsy or surgical resection, based upon the clinical situation. Standard operating procedures for biopsies, sample preparation and analysis have been defined.
Time Frame: Up to 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Dabrafenib and Trametinib
Number analyzed (Participants) | 13
percentage of participants | 92

6. Secondary Outcome: Percentage of Biopsies With Adequate Tissue for Biomarker Analysis
Description: Measured by the percent of tumor necrosis on hematoxylin and eosin stains; RNA gel electrophoresis, percent of adequate tissue for immunohistochemical stains in tissue microarray and cyTOF analysis.
Time Frame: Up to 3 months
Measure: Number; unit: percentage of biopsies w/adequate tissue
Arm/Group | Dabrafenib and Trametinib
Number analyzed (Participants) | 13
percentage of biopsies w/adequate tissue | 92

ADVERSE EVENTS:
Time Frame: Serious adverse events and Adverse events were collected over 25 months period.
Arm/Group | Basic Science (Dabrafenib, Trametinib)
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basic Science (Dabrafenib, Trametinib) (N=13)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Kidney Injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basic Science (Dabrafenib, Trametinib) (N=13)
Fatigue (General disorders) | 8 (10)
Chills (General disorders) | 5 (7)
Fever (General disorders) | 3 (4)
Pain (General disorders) | 2 (2)
Edema, limbs (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Generalized skin senstivity (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3)
Lymphocyte count decreased (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Other (Investigations) | 1 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Constipationi (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Other (Cardiac disorders) | 1 (1)
Wound infection (Infections and infestations) | 2 (3)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes